CLINICAL TRIAL: NCT00451958
Title: An Open-Label, Multi-Centre, Extension Study, Evaluating the Long-Term Safety and Tolerability of Degarelix One-Month Dosing Regimen in Patients With Prostate Cancer Requiring Androgen Ablation Therapy
Brief Title: A Long-term Extension Study Evaluating a One-Month Dosing Regimen of Degarelix in Prostate Cancer Requiring Androgen Ablation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS21A; 2006-006913-34 (EudraCT Number)
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Prostate Cancer
Keywords: Degarelix; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Degarelix 80 mg / Degarelix 80 mg (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The subsequent doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections every 28 days for the rest of the study.
  Interventions: Drug: Degarelix 80 mg / Degarelix 80 mg
- Degarelix 160 mg / Degarelix 160 mg (Experimental): The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 as two 3 mL subcutaneous (s.c.) injections. The subsequent monthly degarelix maintenance dose of 160 mg (40 mg/mL) degarelix were administered as single 4 mL s.c. injections every 28 days.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
  Interventions: Drug: Degarelix 160 mg / Degarelix 160 mg
- Leuprolide 7.5 mg / Degarelix 80 mg (Experimental): During the main CS21 study, leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
  Interventions: Drug: Leuprolide 7.5 mg / Degarelix 80 mg
- Leuprolide 7.5 mg / Degarelix 160 mg (Experimental): During the main CS21 study, leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
  Interventions: Drug: Leuprolide 7.5 mg / Degarelix 160 mg

INTERVENTIONS:
Drug: Degarelix 80 mg / Degarelix 80 mg
  Other Names: Firmagon
  Arms: Degarelix 80 mg / Degarelix 80 mg
Drug: Degarelix 160 mg / Degarelix 160 mg
  Other Names: Firmagon
  Arms: Degarelix 160 mg / Degarelix 160 mg
Drug: Leuprolide 7.5 mg / Degarelix 80 mg
  Other Names: Firmagon; Lupron
  Arms: Leuprolide 7.5 mg / Degarelix 80 mg
Drug: Leuprolide 7.5 mg / Degarelix 160 mg
  Other Names: Firmagon; Lupron
  Arms: Leuprolide 7.5 mg / Degarelix 160 mg

SUMMARY:
Participants who completed the FE200486 CS21 study (NCT00295750) could enter the FE200486 CS21A study. The study continued until all non-discontinued participants had received treatment for at least 5 years.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Patients with histologically proven prostate cancer of all stages in whom endocrine treatment is indicated.
* Signed informed consent
* The patients must have completed the FE 200486 CS21 Study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2007-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (69):
- United States (14):
  - Urology Centers Of Alabama, Homewood, Alabama
  - South Orange County Medical Research Center, Laguna Hills, California
  - Western Clinical Research, Torrance, California
  - Urology Associates Research, Englewood, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Investigational Site, Ocala, Florida
  - Regional Urology, Shreveport, Louisiana
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Investigational Site, Carmel, New York
  - North Urology Research, Concord, North Carolina
  - Investigational Site, Greensboro, North Carolina
  - State College Urologic Association, State College, Pennsylvania
  - Urology San Antonio Research, San Antonio, Texas
  - Seattle Urology Research Center, Burien, Washington
- Canada (9):
  - Investigational Site, Kentville, Nova Scotia
  - The Female/Male Health Centres, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - Burlington Professional Centre, Burlington, Ontario
  - The Urology Research Centre, Burlington, Ontario
  - Investigational Site, Newmarket, Ontario
  - The Female/Male Health Centres, Oakville, Ontario
  - Urology South Shore Research, Greenfields, Quebec
  - Can-Med Clinical Research Inc, Victoria
- Czechia (7):
  - Urocentrum Brno, Brno
  - UROHELP - Bozetechova, Brno
  - Nemocnice Jindrichuv Hradec, a.s., Jindřichův Hradec
  - Fakultni Nemocnice Olomouc, Olomouc
  - Slezska nemocnice, Opava
  - Fakultni nemocnice v Motole, Prague5, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague2, Prague
- Germany (2):
  - Klinikum Mannheim Universitätsklinikum GmbH, Mannheim
  - Klinikum der Universität Regensburg, Regensburg
- Hungary (7):
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Dombóvári Szent Lukács Egészségügyi Kht., Dombóvár
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Miskolci Semmelweis Ignác Egészségügyi Központ és Egyetemi Oktató Kórház Nonprofit Kft, Miskolc
  - Pécsi Tudományegyetem, Pécs
  - Investigational Site, Szeged
- Mexico (8):
  - Investigational Site, Acapulco
  - Hospital Christus Muguerza del Parque, Chihuahua, Chih.
  - Investigational Sit, Durango
  - Hospital Aranda de la Parra , S.A. de C.V., Leon, GTO
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran Mexico, DF Mexico, Mexico City
  - Investigational Site, Mexico City
  - Consultorio Medico, Zapopan, Jalisco
  - Investigational Site, Zapopan, Jalisco
- Netherlands (3):
  - Investigational Site, Ede
  - Investigational Site, Eindhoven
  - Atrium MC, Heerlen
- Hospital Andres Grillasca, Ponce, Puerto Rico
- Romania (7):
  - Investigational Site, Arad
  - Fundeni Uronephrology and Renal Transplant Clinical Institute, Bucharest
  - Investigational Site, Bucharest
  - Sfantul Ioan" Emergency Clinical Hospital, Bucharest
  - PROVITA 2000 Medical Center, Constanța
  - Investigational Site, Iași
  - Sibiu Emergency Clinical County Hospital, Sibiu
- Russia (6):
  - City Clinical Hospital #1 n.a. N.I.Pirogov, Moscow
  - City Clinical Hospital #60, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - City Pokrovskaya Hospital, Saint Petersburg
  - Investigational Site, Saint Petersburg
  - St.Petersburg State Medical Academy n. a. I.I.Mechnikov, Saint Petersburg
- Ukraine (4):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Regional Clinical Center of Urology and Nephrology n.a. V.I.Shapoval, Kharkiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Odesa State Medical University, Odesa
- Clatterbridge Centre For Oncology, Bebington, Wirral, United Kingdom

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants who completed the CS21 study (NCT00295750) were eligible to enrol into the CS21A extension study. Since the number of participants who completed this long-term study was low, no firm conclusions can be drawn from the results.
Pre-assignment Details: Initially, participants treated with degarelix during CS21 continued to treatment and patients who received treatment with leuprolide during CS21 were re-randomised to one of the two degarelix treatment regimens. Following a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg for the rest of the study.
Groups:
- Degarelix 80 mg / Degarelix 80 mg: The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 of the CS21 study (NCT00295750) as two 3 mL subcutaneous (s.c.) injections. The subsequent doses of 80 mg (20 mg/mL) degarelix were administered as single 4 mL s.c. injections every 28 days for the rest of the CS21 study and the current CS21A study.
- Degarelix 160 mg / Degarelix 160 mg: The degarelix doses were administered into the abdominal wall every 28 days. A starting dose of 240 mg (40 mg/mL) degarelix was administered on Day 0 of the CS21 study (NCT00295750) as two 3 mL subcutaneous (s.c.) injections. The subsequent monthly degarelix maintenance dose of 160 mg (40 mg/mL) degarelix were administered as single 4 mL s.c. injections every 28 days for the rest of the CS21 study and the current CS21A study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
- Leuprolide 7.5 mg / Degarelix 80 mg; Leuprolide 7.5 mg / Degarelix 160 mg: During the main CS21 study (NCT00295750), leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
- Leuprolide 7.5 mg: During the main CS21 study (NCT00295750), leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  When the main CS21 study was completed these patients were switched to treatment with degarelix 80 mg or 160 mg in the CS21A study.
Period: CS21 (NCT00295750)
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg | Leuprolide 7.5 mg
Started | 210 (CS21 intention-to-treat (ITT) population.) | 206 (CS21 ITT population.) | 0 (Participants were switched from the leuprolide 7.5 mg group when CS21 was completed.) | 0 (Participants were switched from the leuprolide 7.5 mg group when CS21 was completed.) | 204
Completed | 169 | 163 | 0 | 0 | 172
Not Completed | 41 | 43 | 0 | 0 | 32
Period: CS21A (NCT00451958)
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg | Leuprolide 7.5 mg
Started | 125 (CS21A intention-to-treat (ITT) population.) | 126 (CS21A ITT population.) | 69 (CS21A ITT population.) | 66 (One of the enrolled participants never received any treatment, i.e. the CS21A ITT population=65.) | 0 (Participants were switched to the degarelix groups when CS21 was completed.)
Completed | 60 | 49 | 27 | 27 | 0
Not Completed | 65 | 77 | 42 | 39 | 0
Not completed — Adverse Event | 21 | 34 | 14 | 17 | 0
Not completed — Lost to Follow-up | 6 | 5 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 3 | 2 | 0 | 0
Not completed — Physician Decision | 2 | 4 | 4 | 4 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 4 | 3 | 0
Not completed — Miscellaneous reasons | 28 | 27 | 17 | 14 | 0

BASELINE CHARACTERISTICS:
Population: CS21A intention-to-treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg | Total
Number analyzed (Participants) | 125 | 126 | 69 | 65 | 385
Age Continuous [Mean (Standard Deviation); unit: years] — CS21A intention-to-treat (ITT) population.
  years | 70.1 (7.62) | 71.1 (8.25) | 72.4 (9.46) | 71.4 (8.24) | 71.1 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants] — CS21A ITT population.
  Participants
    Female | 0 | 0 | 0 | 0 | 0
    Male | 125 | 126 | 69 | 65 | 385
Region of Enrollment [Number; unit: participants] — CS21A ITT population.
  participants
    United States | 12 | 14 | 13 | 9 | 48
    Hungary | 7 | 9 | 5 | 5 | 26
    Czech Republic | 11 | 12 | 6 | 8 | 37
    Mexico | 15 | 17 | 10 | 7 | 49
    Canada | 4 | 5 | 5 | 4 | 18
    Ukraine | 11 | 10 | 7 | 3 | 31
    Romania | 36 | 39 | 16 | 15 | 106
    Russian Federation | 26 | 19 | 6 | 13 | 64
    Netherlands | 2 | 0 | 0 | 1 | 3
    Germany | 0 | 0 | 1 | 0 | 1
    United Kingdom | 1 | 1 | 0 | 0 | 2
Body Weight [Mean (Standard Deviation); unit: kilogram] — CS21A ITT population.
  kilogram | 78.4 (12.6) | 79.2 (13.4) | 78.7 (11.3) | 80.0 (12.1) | 79.0 (12.5)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] — CS21A ITT population.
  kilogram per square meter | 26.4 (3.92) | 26.9 (3.79) | 26.9 (3.94) | 27.1 (3.67) | 26.8 (3.84)
Gleason Score [Number; unit: participants] — CS21A ITT population. The Gleason Score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive. Two of the participants did not have a Gleason Score at Baseline.
  participants
    Gleason Score 2-4 | 15 | 17 | 8 | 11 | 51
    Gleason Score 5-6 | 37 | 44 | 25 | 18 | 124
    Gleason Score 7-10 | 73 | 63 | 36 | 36 | 208
Stage of Prostate Cancer [Number; unit: participants] — CS21A ITT population. Prostate cancer stage was classified according to the Tumor, Nodes, and Metastatic (TNM) scale to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localised | 39 | 36 | 20 | 19 | 114
    Locally advanced | 46 | 44 | 18 | 24 | 132
    Metastatic | 23 | 22 | 21 | 9 | 75
    Not classifiable | 17 | 24 | 10 | 13 | 64
Serum Testosterone Levels [Median (Full Range); unit: nanograms per milliliter] — CS21A ITT population.
  nanograms per milliliter | 4.63 [1.28 to 10.6] | 4.02 [0.55 to 10.6] | 4.32 [1.34 to 12.5] | 3.51 [0.37 to 8.00] | 4.23 [0.37 to 12.5]
Serum Prostate-Specific Antigen (PSA) Levels [Median (Full Range); unit: nanograms per milliliter] — CS21A ITT population.
  nanograms per milliliter | 22.2 [1.70 to 3187] | 22.5 [1.50 to 4902] | 25.5 [1.60 to 2112] | 14.0 [1.60 to 10952] | 21.0 [1.50 to 10952]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Markedly Abnormal Values in Vital Signs and Body Weight
Description: This outcome measure included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight. The table presents the number of participants with normal baseline (from main CS21 study, NCT00295750) and at least one post-baseline markedly abnormal value during CS21A.
Time Frame: Up to 4 years of treatment
Population: The analysis population comprised all participants who were enrolled in the CS21A study and who received at least one dose of degarelix during the study period.
Measure: Number; unit: participants
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg
Number analyzed (Participants) | 125 | 126 | 69 | 66
participants
  Diastolic blood pressure <=50 and decrease >=15 | 3 | 6 | 3 | 6
  Diastolic blood pressure >=105 and increase >=15 | 3 | 6 | 4 | 0
  Systolic blood pressure <=90 and decrease >=20 | 4 | 4 | 5 | 3
  Systolic blood pressure >=180 and increase >=20 | 7 | 13 | 7 | 4
  Heart rate <=50 and decrease >=15 | 4 | 3 | 7 | 2
  Heart rate >=120 and increase >=15 | 1 | 1 | 1 | 3
  Body weight decrease of >=7 percent | 15 | 24 | 21 | 8
  Body weight increase of >=7 percent | 25 | 14 | 4 | 5

2. Primary Outcome: Number of Participants With Markedly Abnormal Values in Safety Laboratory Variables
Description: This outcome measure included incidence of markedly abnormal changes in safety laboratory values. The table presents the number of participants with normal baseline (from main CS21 trial, NCT00295750) and at least one post-baseline markedly abnormal value during CS21A. Only the laboratory variables that had at least five percentages of participants in either group with abnormal value are presented, more variables were included in the study. ULN=Upper limit of normal.
Time Frame: Up to 4 years of treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg
Number analyzed (Participants) | 125 | 126 | 69 | 65
participants
  S-Potassium (mmol/L) >=5.8 | 11 | 9 | 6 | 5
  S-Alanine aminotransferase (IU/L) >3xULN | 1 | 6 | 1 | 0
  S-Alkaline phosphatase (IU/L) >3xULN+25% increase | 4 | 5 | 4 | 2
  S-Creatinine (µmol/L) >=177 | 12 | 7 | 5 | 2
  S-Urea nitrogen (mmol/L) >=10.7 | 6 | 9 | 5 | 5
  B-Haematocrit (Ratio) <=0.37 | 40 | 47 | 22 | 17
  B-Haemoglobin (g/L) <=115 | 12 | 20 | 9 | 6
  B-Red blood cell count (10^12/L) <=3.5 | 10 | 15 | 5 | 3
  B-Eosinophils (%) >=10 | 6 | 7 | 1 | 1
  B-Lymphocytes (%) <=10 | 8 | 9 | 10 | 5

3. Secondary Outcome: Percentage of Participants With no Prostate-specific Antigen (PSA) Progression
Description: PSA progression was defined as two consecutive increases of 50%, and at least 5 ng/mL, compared to nadir (obtained in either CS21, NCT00295750, or CS21A). The figures below present the percentage of participants with no PSA progression at each of the selected time points (there were more time points in the study) along with corresponding 95% confidence intervals (CI).
Time Frame: Until all participants have received at least 5 years of treatment and at a frequency of every 3 months
Population: CS21 ITT analysis set i.e. all participants who received at least one dose of degarelix or leuprolide during the mail study (CS21).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg
Number analyzed (Participants) | 207 | 202 | 69 | 132
percentage of participants
  Day 28 | 100 [100 to 100] | 99.5 [96.5 to 99.9] | 98.6 [90.2 to 99.8] | 100 [100 to 100]
  Day 364 | 91.1 [85.9 to 94.5] | 85.8 [79.8 to 90.1] | 82.6 [71.4 to 89.7] | 87.9 [80.4 to 92.7]
  Day 1960 | 61.0 [50.9 to 69.7] | 58.7 [48.7 to 67.4] | 50.7 [36.3 to 63.4] | 73.8 [60.9 to 83.0]

4. Secondary Outcome: Percentage of Participants With Testosterone Level Maintained at <=0.5 ng/mL From Day 28 in CS21 and Onwards
Description: The results below present the percentage of participants of having testosterone <=0.5 ng/mL at each of the selected time points (there were more time points in the study) from Day 28 in CS21 (NCT00295750) until the end of the CS21A study.
  In all treatment groups approximately 3% per year of the participants had at least one testosterone >0.5 ng/mL during the study.
Time Frame: Until all participants have received at least 5 years of treatment and at a frequency of every 6 months
Population: CS21 ITT analysis set i.e. all participants who received at least one dose of degarelix or leuprolide during the mail CS21 study (NCT00295750).
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Leuprolide 7.5 mg / Degarelix 160 mg: During the main CS21 study, leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Leuprolide participants who dropped out during the first year (i.e. during CS21) were all attributed to what became the leuprolide 7.5 mg / degarelix 160 mg arm.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg
Number analyzed (Participants) | 206 | 197 | 69 | 128
percentage
  Day 84 | 99.5 [96.5 to 99.9] | 100 [100 to 100] | 98.6 [90.2 to 99.8] | 97.6 [92.7 to 99.2]
  Day 364 | 97.2 [93.5 to 98.8] | 98.3 [94.8 to 99.4] | 97. [88.9 to 99.3] | 96.0 [90.5 to 98.3]
  Day 1876 | 82.0 [72.7 to 88.4] | 87.7 [78.0 to 93.3] | 84.1 [70.2 to 91.9] | 88.4 [75.5 to 94.7]

5. Secondary Outcome: Serum Levels of Testosterone From the Time of Switch From Leuprolide to Degarelix up to Day 56
Time Frame: From time of switch to Day 56
Population: All participants who received leuprolide in the main CS21 study (NCT00295750) and were switched over to degarelix in the CS21A extension study.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Leuprolide 7.5 mg/ Degarelix 240/80 mg: During the main CS21 study (NCT00295750), leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
- Leuprolide 7.5 mg/ Degarelix 240/160 mg: During the main CS21 study, leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
Arm/Group | Leuprolide 7.5 mg/ Degarelix 240/80 mg | Leuprolide 7.5 mg/ Degarelix 240/160 mg
Number analyzed (Participants) | 69 | 64
ng/mL
  Baseline | 0.076 [0.015 to 1.36] | 0.074 [0.015 to 0.229]
  Day 3 | 0.084 [0.015 to 0.23] | 0.068 [0.015 to 0.19]
  Day 7 | 0.076 [0.015 to 0.22] | 0.066 [0.015 to 0.16]
  Day 14 | 0.085 [0.015 to 0.24] | 0.073 [0.015 to 0.27]
  Day 28 | 0.074 [0.015 to 0.21] | 0.074 [0.015 to 0.19]
  Day 56 | 0.080 [0.015 to 0.22] | 0.077 [0.015 to 0.16]

6. Secondary Outcome: Serum Levels of PSA From the Time of Switch From Leuprolide to Degarelix to Day 56
Time Frame: From time of switch to Day 56
Population: as for outcome 5
Measure: Median (Full Range); unit: ng/mL
Groups:
- Leuprolide 7.5 mg/ Degarelix 240/80 mg; Leuprolide 7.5 mg/ Degarelix 240/160 mg: During the main CS21 study, leuprolide (Lupron Depot) 7.5 mg was injected into the muscle every 28 days for one year.
  Starting one year after the first dose of leuprolide, degarelix doses were administered into the abdominal wall every 28 days. First, a starting dose of 240 mg (40 mg/mL) degarelix was administered as two 3 mL subcutaneous (s.c.) injections and one month later the participants received either subsequent monthly degarelix maintenance doses of 80 mg (20 mg/mL) or 160 mg (40 mg/mL) every 28 days for the rest of the study.
  Following the implementation of a protocol amendment, all patients received a monthly degarelix maintenance dose of 80 mg (20 mg/mL) for the rest of the study.
Arm/Group | Leuprolide 7.5 mg/ Degarelix 240/80 mg | Leuprolide 7.5 mg/ Degarelix 240/160 mg
Number analyzed (Participants) | 69 | 65
ng/mL
  Baseline | 0.4 [0 to 2938] | 0.4 [0 to 1096]
  Day 3 | 0.4 [0 to 754] | 0.3 [0 to 1059]
  Day 7 | 0.35 [0 to 724] | 0.4 [0 to 1422]
  Day 14 | 0.4 [0 to 671] | 0.3 [0 to 1567]
  Day 28 | 0.4 [0 to 441] | 0.5 [0 to 2008]
  Day 56 | 0.35 [0 to 620] | 0.4 [0 to 1926]

7. Secondary Outcome: Serum Levels of Luteinizing Hormone (LH) From the Time of Switch From Leuprolide to Degarelix to Day 56
Time Frame: From time of switch to Day 56
Population: as for outcome 5
Measure: Median (Full Range); unit: International units/Liter (IU/L)
Arm/Group | Leuprolide 7.5 mg/ Degarelix 240/80 mg | Leuprolide 7.5 mg/ Degarelix 240/160 mg
Number analyzed (Participants) | 69 | 65
International units/Liter (IU/L)
  Baseline | 0.035 [0.035 to 1.12] | 0.035 [0.035 to 0.40]
  Day 3 | 0.035 [0.035 to 0.11] | 0.035 [0.035 to 0.12]
  Day 7 | 0.035 [0.035 to 0.11] | 0.035 [0.035 to 0.08]
  Day 14 | 0.035 [0.035 to 0.47] | 0.035 [0.035 to 0.12]
  Day 28 | 0.035 [0.035 to 0.16] | 0.035 [0.035 to 0.19]
  Day 56 | 0.035 [0.035 to 0.17] | 0.035 [0.035 to 0.22]

8. Secondary Outcome: Serum Levels of Follicle Stimulating Hormone (FSH) From the Time of Switch From Leuprolide to Degarelix to Day 56
Time Frame: From time of switch to Day 56
Population: as for outcome 5
Measure: Median (Full Range); unit: International units/Liter (IU/L)
Arm/Group | Leuprolide 7.5 mg/ Degarelix 240/80 mg | Leuprolide 7.5 mg/ Degarelix 240/160 mg
Number analyzed (Participants) | 69 | 65
International units/Liter (IU/L)
  Baseline | 4.8 [1.2 to 15.8] | 4.4 [1.5 to 12.2]
  Day 3 | 2.7 [0.8 to 11.1] | 2.8 [0.5 to 7.6]
  Day 7 | 2.6 [0.7 to 11.8] | 2.6 [0.4 to 6.9]
  Day 14 | 2.2 [0.15 to 7.9] | 2.3 [0.15 to 8.3]
  Day 28 | 1.8 [0.15 to 7.6] | 1.7 [0.15 to 6.7]
  Day 56 | 1.3 [0.15 to 6.7] | 1.55 [0.15 to 5.6]

ADVERSE EVENTS:
Time Frame: From start of CS21A and up to 4.5 years.
Description: The population comprised all participants who were enrolled into CS21A and who received at least one dose of degarelix during the study.
Arm/Group | Degarelix 80 mg / Degarelix 80 mg | Degarelix 160 mg / Degarelix 160 mg | Leuprolide 7.5 mg / Degarelix 80 mg | Leuprolide 7.5 mg / Degarelix 160 mg
Serious Adverse Events (participants affected / at risk) | 43/207 | 60/202 | 23/69 | 22/66
Other Adverse Events (participants affected / at risk) | 181/207 | 177/202 | 63/69 | 58/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 80 mg / Degarelix 80 mg (N=207) | Degarelix 160 mg / Degarelix 160 mg (N=202) | Leuprolide 7.5 mg / Degarelix 80 mg (N=69) | Leuprolide 7.5 mg / Degarelix 160 mg (N=66)
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 1 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 2 | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Accidental death (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal gangrene (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to biliary tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Non-hodgkin's lymphoma unspecified histology indolent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamus cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 2 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 6 | 2 | 2
Calculus bladder (Renal and urinary disorders) | 2 | 1 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 3 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 2 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Myopericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia obstructive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
ECG signs of myocardial ischaemia (Investigations) | 0 | 0 | 0 | 1
Prostate examination abnormal (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Malignant lymphoma unclassifiable high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pleural mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0
Hyperkinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Squamus cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 80 mg / Degarelix 80 mg (N=207) | Degarelix 160 mg / Degarelix 160 mg (N=202) | Leuprolide 7.5 mg / Degarelix 80 mg (N=69) | Leuprolide 7.5 mg / Degarelix 160 mg (N=66)
Anaemia (Blood and lymphatic system disorders) | 17 | 18 | 10 | 6
Atrial fibrillation (Cardiac disorders) | 2 | 6 | 4 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 4 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 17 | 13 | 12 | 10
Constipation (Gastrointestinal disorders) | 18 | 12 | 9 | 2
Nausea (Gastrointestinal disorders) | 10 | 15 | 3 | 6
Vomiting (Gastrointestinal disorders) | 4 | 7 | 6 | 3
Injection site pain (General disorders) | 65 | 67 | 20 | 16
Injection site erythema (General disorders) | 40 | 51 | 10 | 16
Pyrexia (General disorders) | 20 | 22 | 8 | 9
Injection site swelling (General disorders) | 17 | 16 | 6 | 4
Fatigue (General disorders) | 12 | 15 | 9 | 6
Asthenia (General disorders) | 13 | 13 | 8 | 3
Injection site nodule (General disorders) | 13 | 17 | 4 | 2
Injection site inflammation (General disorders) | 7 | 5 | 6 | 0
Urinary tract infection (Infections and infestations) | 12 | 10 | 14 | 10
Influenza (Infections and infestations) | 12 | 10 | 8 | 2
Nasopharyngitis (Infections and infestations) | 11 | 7 | 5 | 5
Weight decreased (Investigations) | 20 | 24 | 19 | 10
Alanine aminotransferase increased (Investigations) | 19 | 21 | 6 | 6
Prostatic specific antigen increased (Investigations) | 16 | 20 | 10 | 6
Aspartate aminotransferase increased (Investigations) | 15 | 14 | 7 | 5
Gamma-glutamyltransferase increased (Investigations) | 8 | 15 | 7 | 2
Blood creatinine increased (Investigations) | 11 | 9 | 5 | 4
Blood alkaline phosphatase increased (Investigations) | 7 | 11 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 20 | 10 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 14 | 14 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 9 | 7 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 45 | 4 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 11 | 5 | 6
Dizziness (Nervous system disorders) | 13 | 14 | 5 | 6
Headache (Nervous system disorders) | 11 | 10 | 5 | 5
Insomnia (Psychiatric disorders) | 10 | 9 | 2 | 8
Depression (Psychiatric disorders) | 3 | 11 | 4 | 6
Urinary retention (Renal and urinary disorders) | 5 | 14 | 7 | 6
Haematuria (Renal and urinary disorders) | 10 | 11 | 4 | 3
Dysuria (Renal and urinary disorders) | 5 | 11 | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 5 | 2
Hot flush (Vascular disorders) | 62 | 63 | 20 | 21
Hypertension (Vascular disorders) | 19 | 27 | 8 | 5
Myocardial infarction (Cardiac disorders) | 4 | 2 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 8 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 5 | 4 | 0
Chest pain (General disorders) | 2 | 3 | 4 | 0
Chills (General disorders) | 16 | 11 | 3 | 2
Injection site induration (General disorders) | 9 | 13 | 1 | 3
Oedema peripheral (General disorders) | 8 | 9 | 4 | 3
Bronchitis (Infections and infestations) | 8 | 6 | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 5 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 8 | 4 | 0
Blood urea increased (Investigations) | 9 | 5 | 4 | 0
Weight increased (Investigations) | 32 | 25 | 15 | 14
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 18 | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 1 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 7 | 2 | 4
Calculus ureteric (Renal and urinary disorders) | 2 | 0 | 0 | 3
Cystitis noninfective (Renal and urinary disorders) | 2 | 2 | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 3 | 5 | 2 | 4
Nocturia (Renal and urinary disorders) | 6 | 4 | 2 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 4 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.